## Statistical Analysis Plan for Part I and Part II

**Title:** A phase I, open-label, fixed-sequence, single-center study to determine the effect of repeated dosing with clarithromycin on the pharmacokinetics of linaprazan glurate/linaprazan and the effect of a single dose of linaprazan glurate on the pharmacokinetics of clarithromycin, and single and repeated dosing with linaprazan glurate on the pharmacokinetics of midazolam administrated to healthy subjects

NCT number: NCT05633147

**Document date:** Final v1.0; 06MAR2023



# Statistical Analysis Plan for Part I and Part II

EudraCT no. 2022-001403-41

Investigational medicinal product Linaprazan glurate

Study code CX842A2105

Protocol version and date Final v4.0; 20JAN2023

A phase I, open-label, fixed-sequence, single-center study to determine the effect of repeated dosing with clarithromycin on the pharmacokinetics of linaprazan glurate/linaprazan and the effect of a single dose of linaprazan glurate on the pharmacokinetics of clarithromycin, and single and repeated dosing with linaprazan glurate on the pharmacokinetics of midazolam administrated to healthy subjects

Sponsor signatory , MD, PhD, CMO

Cinclus Pharma Holding AB World Trade Center, Kungsbron 1 SE-111 22 Stockholm, Sweden

CTC biostatistician, MSc

Clinical Trial Consultants AB (CTC) Dag Hammarskjölds väg 10B SE-752 37 Uppsala, Sweden

This Statistical Analysis Plan is the property of Cinclus Pharma Holding AB and is a confidential document. It is not to be copied or distributed to other parties without written approval from Cinclus Pharma Holding AB.




#### 1 SIGNATURES

## Author of this statistical analysis plan (SAP)



## Sponsor representative signatory



## Sponsor biostatistician signatory






## 2 TABLE OF CONTENTS

| 1 | SIG | NATURES | 2 |
|---|------------|-------------------------------------------------|------|
| 2 | TAI | BLE OF CONTENTS | 3 |
| 3 | LIS | T OF ABBREVIATIONS AND DEFINITION OF TERMS | 5 |
| 4 | INT | RODUCTION | 7 |
| | 4.1 | Study design | 7 |
| | 4.2 | Study objectives and endpoints Part I | 7 |
| | 4.3 | Study objectives and endpoints Part II | 8 |
| | 4. | 3.1.1 Additional PK parameters Part II | 9 |
| | 4.4 | Randomisation and number of subjects | . 10 |
| | 4.5 | Subject replacement | . 10 |
| | 4.6 | Blinding | . 10 |
| 5 | STA | ATISTICAL AND ANALYTICAL PLANS | . 11 |
| | 5.1 | Statistical hypotheses | . 11 |
| | 5.2 | Sample size calculation | . 11 |
| | 5.3 | Definition of analysis sets | . 11 |
| | <b>5.4</b> | Compliance | . 11 |
| | 5.5 | Definition of baseline | . 12 |
| | 5.6 | Rounding principles | . 12 |
| | <b>5.7</b> | Significance level | |
| | 5.8 | Multiple comparisons/multiplicity | |
| | 5.9 | Handling of dropouts, missing data and outliers | |
| 6 | | ANGES FROM THE CLINICAL STUDY PROTOCOL | |
| 7 | CLI | NICAL DATABASE PROCESSING | |
| | 7.1 | General information | . 15 |
| | 7.1. | CDISC Compliance | . 15 |
| | 7.2 | Database modeling of study design | |
| 8 | | TISTICAL DELIVERABLES | |
| 9 | STA | TISTICAL METHODOLOGY | |
| | 9.1 | Pharmacokinetic calculations | |
| | 9.2 | Analysis of the primary endpoint | . 21 |
| | 9.2. | | |
| | 9.2.2 | 1 | |
| | 9.2.3 | Mixed model for PK parameters Part II | . 22 |
| | 9.3 | Analysis of secondary endpoints | |
| | 9.3. | Adverse events | . 22 |

| 1 | Cınclı | us Pharma | |
|---|---|---|---|
| | | Statistical Analysis Plan for Part I and Part II CX842A2105 FINAL v | |
| | 9.3.2 | Physical examinations. | |
| | 9.3.3 | Vital signs | |
| | 9.3.4 | 12-lead safety ECG | . 22 |
| | 9.3.5 | Safety laboratory analyses | . 22 |
| | 9.3.6 limited | Additional PK parameters Part I for linaprazan glurate and linaprazan, not to: | . 22 |
| | 9.3.7<br>linapraz | Clarithromycin PK parameters Part I with and without co-administration of an glurate: | . 23 |
| | 9.3.8<br>linapraz | Additional Midazolam PK parameters Part II in the presence and absence of an glurate administration (if feasible): | . 23 |
| | 9.3.9 | Linaprazan glurate and linaprazan PK parameters Part II (if feasible): | . 23 |
| 9. | 4 De | scription of study population | . 23 |
| 10 | DATA 1 | DISPLAY PLAN | . 24 |
| 1( | 0.1 Ta | ble of contents DDP | . 24 |
| Lis | t of table | es | |
| Tabl | le 1 | Analysis sets | 11 |
| List | of figur | es | |
| Figu | ıre 1 | Schematic representation of the SDTM study design | 16 |




## 3 LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation | Explanation |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse event |
| ATC | Anatomical therapeutic chemical |
| AUC | Area under the plasma concentration vs. time curve |
| $\mathrm{AUC}_{0	ext{-t}}$ | AUC from time 0 to time t |
| AUC <sub>extr%</sub> | AUC percent extrapolation |
| AUCinf | AUC from 0 to infinity |
| AUC <sub>tau</sub> | AUC to end of dosing period |
| BID | Bis in die, twice daily |
| CDISC | Clinical Data Interchange Standards Consortium |
| CF | Clean File |
| CI | Confidence interval |
| CL | Apparent total body clearance following i.v. administration |
| CL/F | Apparent total body clearance following extravascular administration |
| $C_{last}$ | Last observed plasma concentration |
| $C_{\text{max}}$ | Maximum observed concentration |
| CS | Clinically significant |
| CSP | Clinical study protocol |
| CSR | Clinical study report |
| CT | Controlled terminology |
| CTC | Clinical Trial Consultants AB |
| CV | Coefficient of variation |
| DDI | Drug-drug interaction |
| DDP | Data display plan |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| FAS | Full analysis set |
| FDA | United States Food and Drug Administration |
| Geo | Geometric |
| IG | Implementation guideline |
| IMP | Investigational medicinal product |
| lin | Linear |




Statistical Analysis Plan for Part I and Part II CX842A2105 FINAL v1.0

## **Abbreviation** Explanation

LLOQ Lower limit of quantification

LS Least square
Max Maximum

Medical dictionary for regulatory activities

Min Minimum

NA Not applicable/not available

NC Not calculated

NCA Non-compartmental analysis

NCS Not clinically significant

PgP P-glycoprotein

PK Pharmacokinetic(s)

PKAS PK analysis set

PT Preferred term

R<sub>acc</sub> Accumulation ratio

SAE Serious adverse event

SAP Statistical analysis plan

SD Standard deviation

SDTM Study data tabulation model

SOC System organ class

 $T_{last} \hspace{1cm} Time \ of \ occurrence \ of \ C_{last} \\ T_{max} \hspace{1cm} Time \ of \ occurrence \ of \ C_{max}$ 

T<sub>1/2</sub> Terminal elimination half-life

V/F Volume of distribution following extravascular

administration




#### 4 INTRODUCTION

## 4.1 Study design

This is a phase I, open-label, fixed design, drug-drug-interaction (DDI) study divided in 2 parts. Part I is designed to evaluate whether concomitant treatment with linaprazan glurate and clarithromycin, a strong inhibitor of cytochrome P450 3A4 (CYP3A4) and P-glycoprotein P (PgP), leads to an effect on the systemic exposure to linaprazan glurate and linaprazan and whether there is an effect on the pharmacokinetics of clarithromycin after a single dose of linaprazan glurate. Part II is designed to evaluate the effect of repeated doses of linaprazan glurate on the pharmacokinetics (PK) of a sensitive substrate of CYP3A (midazolam).

For more details on the study design, please refer to the CSP.

## 4.2 Study objectives and endpoints Part I

| Objectives | Endpoints | Assessments | Analyses | Data display<br>plan (DDP) |
|---|---|---|---|---|
| Primary<br>objective,<br>Part I | Primary endpoint,<br>Part I | Assessments, Part I | Analyse, Part I | DDP, Part I |
| To investigate the effect of repeated administration of clarithromycin on linaprazan glurate and linaprazan PK after single dose of linaprazan glurate. | Linaprazan glurate and linaprazan PK parameters with and without co-administration of clarithromycin: Area under the plasma concentration curve from 0 to infinity (AUC <sub>inf</sub> ) AUC from time 0 to time t (AUC <sub>0-t</sub> ) Maximum plasma concentration (C <sub>max</sub> ) | Pharmacokinetic sampling and analysis | Summary statistics for PK parameters. See Section 9. Linear mixed-effects analysis of variance model, see Section 9.2.2 | Table PP 1, Table PC 1 and Figure PC 1 |
| Secondary<br>objective,<br>Part I | Secondary endpoint,<br>Part I | Assessments, Part I | Analyse, Part I | DDP, Part I |
| To assess the safety and tolerability | Frequency, seriousness, and intensity of AEs. | Adverse events | Descriptive statistics,<br>Section 9.3.1 | Table AE 1,<br>Table AE 3 |
| after single<br>dose of<br>linaprazan<br>glurate with<br>and without<br>co-<br>administration<br>of<br>clarithromycin. | Clinically significant changes in physical examinations, vital signs (blood pressure and pulse), electrocardiograms (ECG), and laboratory variables (haematology, clinical chemistry, and urinalysis). | Physical examinations,<br>Vital signs, 12-lead<br>electrocardiograms, Safety<br>laboratory assessments | Descriptive statistics,<br>Section 9.3.2 to 9.3.5 | Table PE 1, Table VS 1, Table EG 1, Table EG 3, Table LB 1, Table LB 3 and Table LB 5 |
| To evaluate additional PK characteristics | Additional PK parameters for linaprazan glurate and | Pharmacokinetic sampling and analysis | Summary statistics for PK parameters. See Section 9.3.6 | Table PP 5 |




| Objectives | Endpoints | Assessments | Analyses | Data display<br>plan (DDP) |
|---|---|---|---|---|
| of linaprazan glurate and | linaprazan, not limited to: | | | • |
| linaprazan. | Time of occurrence of $C_{max}(T_{max})$ | | | |
| | Terminal elimination half-life (T <sub>1/2</sub> ) | - | | |
| | Apparent clearance (CL/F) | - | | |
| | Apparent volume of distribution (V/F) | - | | |
| | Percent extrapolated AUC (AUC <sub>extr</sub> %) | - | | |
| To investigate<br>the effect of<br>linaprazan<br>glurate on<br>clarithromycin | Clarithromycin PK<br>parameters with and<br>without co-<br>administration of<br>linaprazan glurate: | Pharmacokinetic sampling and analysis | Summary statistics for PK parameters. See Section 9.3.7 | _ |
| PK. | AUC to the end of the dosing period (AUC <sub>tau</sub> ) | - | | |
| | $C_{max}$ | | | |
| | Additional PK parameters for clarithromycin, not limited to: | Pharmacokinetic sampling and analysis | _ | |
| | T <sub>max</sub> | - | | |
| | T <sub>1/2</sub> | - | | |
| Exploratory objective, Part I | Exploratory<br>endpoint, Part I | Assessments, Part I | Analyse, Part I | DDP, Part I |
| To explore the metabolites of linaprazan glurate in plasma with and without co-administration of clarithromycin. | Plasma collected for<br>future exploratory<br>analyses of linaprazan<br>glurate metabolites. | Not covered in the SAP | NA | NA |

# 4.3 Study objectives and endpoints Part II

| Objectives | Endpoints | Assessments | Analyses | Data display plan<br>(DDP) |
|---|---|---|---|---|
| Primary<br>objective,<br>Part II | Primary endpoint,<br>Part II | Assessments, Part II | Analyse, Part II | DDP, Part II |
| To investigate<br>the effects<br>after single<br>and repeated | Midazolam PK<br>parameters in the<br>presence and<br>absence of | Pharmacokinetic sampling and analysis | Summary statistics for PK parameters. See Section 9. | |




| Objectives | Endpoints | Assessments | Analyses | Data display plan<br>(DDP) |
|---|---|---|---|---|
| administration of linaprazan | linaprazan glurate administration: | | Linear mixed-<br>effects analysis of | Table PP 2, |
| glurate on the | AUCinf | <del>-</del> | variance model, | |
| PK properties of midazolam. | AUC0-t | _ | see Section 9.2.3 | |
| | Cmax | | | Table PC 2 and |
| | | | | Figure PC 3 |
| Secondary<br>objective,<br>Part II | Secondary<br>endpoint, Part II | Assessments, Part II | Analyse, Part II | DDP, Part II |
| To assess the safety and tolerability | Frequency, seriousness, and intensity of AEs. | Adverse events | Descriptive statistics, Section 9.3.1 | Table AE 2, Table AE 4 |
| after repeated<br>doses of<br>linaprazan<br>glurate with<br>and without<br>co-<br>administration<br>of midazolam. | Clinically significant changes in physical examinations, vital signs (blood pressure and pulse), ECG, and laboratory variables (haematology, clinical chemistry, and urinalysis). | Physical examinations,<br>Vital signs, 12-lead<br>electrocardiograms,<br>Safety laboratory<br>assessments | Descriptive statistics, Section 9.3.2 to 9.3.5 | Table PE 2, Table VS 2,<br>Table EG 2, Table EG<br>4, Table LB 2, Table LB<br>4, Table LB 6 |
| To evaluate PK data on linaprazan glurate and linaprazan after single and repeated oral doses of linaprazan glurate. | Linaprazan glurate and linaprazan PK parameters after repeated administration of linaprazan glurate twice daily (BID) for 13 days (if feasible): AUC <sub>inf</sub> AUC <sub>0-t</sub> C <sub>max</sub> T <sub>max</sub> T <sub>1/2</sub> AUC <sub>extr%</sub> CL/F V/F Accumulation ratio (R <sub>acc</sub> ). | Pharmacokinetic sampling and analysis | Summary statistics for PK parameters. See Section 9.3.9 | 4.3.1.1 Additional PK parameters Part II Table PP 7 |
| To evaluate additional PK characteristics of midazolam in the presence and absence of linaprazan | Midazolam PK<br>parameters in the<br>presence and<br>absence of<br>linaprazan glurate<br>administration (if<br>feasible): | Pharmacokinetic sampling and analysis | Summary statistics for PK parameters. See Section 9.3.8 | |




| Objectives | Endpoints | Assessments | Analyses | Data display plan<br>(DDP) |
|---|---|---|---|---|
| glurate | $T_{\text{max}}$ | | | |
| administration. | T <sub>1/2</sub> | - | | |
| | AUC <sub>extr</sub> % | - | | |
| | CL/F | - | | |
| | V/F | - | | |
| Exploratory objective, Part II | Exploratory endpoint, Part II | Assessments, Part II | Analyse, Part II | DDP, Part II |
| To explore the metabolites of linaprazan glurate in plasma and urine after single and repeated doses of linaprazan glurate. | Plasma and urine<br>collected for future<br>exploratory analyses<br>of linaprazan glurate<br>metabolites. | Not covered in the SAP | NA | NA |

Cinclus Pharma AB is responsible for analysing the exploratory objectives/endpoints. Results related to exploratory objectives/endpoints in Part I and II will not be reported in the clinical study report (CSR). Therefore, these will not be covered in this SAP.

## 4.4 Randomisation and number of subjects

This is a non-randomized study.

In total, approximately 54 subjects will be screened in the study (27 subjects for each part).

In Part I, a total of 18 healthy subjects are planned to be included for an estimated total of 12 evaluable subjects.

In Part II, a total of 18 healthy subjects are planned to be included for an estimated total of 12 evaluable subjects.

#### 4.5 Subject replacement

Subjects who are prematurely withdrawn from the study for any reason except the occurrence of AEs assessed as possibly or probably related to study treatment may be replaced during the course of the study.

### 4.6 Blinding

This is an open-label study, i.e., the Investigator, study staff and study subjects will know the type of treatment received.




## 5 STATISTICAL AND ANALYTICAL PLANS

## 5.1 Statistical hypotheses

The statistical hypothesis to be tested in Part I is that coadministration of linaprazan glurate + clarithromycin as opposed to linaprazan glurate alone has no effect on CYP3A.

The statistical hypothesis to be tested in Part II is that coadministration of midazolam + linaprazan glurate as opposed to midazolam alone has no effect on CYP3A.

#### 5.2 Sample size calculation

No formal sample size calculation has been performed for this study. The proposed sample size is considered sufficient to provide adequate information to meet the study objectives.

## 5.3 Definition of analysis sets

The analysis sets defined for the study are outlined in Table 1.

Table 1 Analysis sets

| Analysis set | Definition | Use of analysis set |
|---|---|---|
| Full analysis set (FAS) | The full analysis set (FAS) will consist of all subjects who have received at least 1 dose of IMP and who provided at least 1 post-baseline data point. There will be 1 FAS per part. | All objectives/endpoints except PK objectives/endpoints. |
| Pharmacokinetic analysis set (PKAS) | The PK analysis set (PKAS) will consist of all subjects who received at least 1 dose of IMP and provided an evaluable plasma concentration profile, and who have no AEs or protocol deviations judged to affect the PK analysis. There will be 1 PKAS per part. Subjects with a calculated compliance of less than 82% during the home administration period will be excluded from the PKAS for the corresponding study part. Individual PK values may be excluded from the analysis as specified in the SAP. All protocol violations will be judged as major or minor prior to database lock. | All PK objectives/endpoints. |

## 5.4 Compliance

During visits at the clinic, the study drugs will be administered at the clinic under medical supervision. Doses administered at the clinic will be entered in the eCRF by study personnel. On other days, subjects will self-administer clarithromycin (Part I) or linaprazan glurate (Part II) at home and register each intake of study drug in an electronic diary. Text reminders will be




sent to the subjects each day. At the compliance visit to the clinic, subjects will be asked to return any unused study drugs and all empty containers.

Percent compliance will be calculated, per study part, for the home administration period as

100 \* (number of tablets delivered – number of tablets returned) / expected number of tablets taken

If the electronic diary indicates the morning dose being taken later than 12.00 or the evening dose being taken before 17.00, the corresponding tablet will be judged as "returned" in the formula above. Calculated percent compliance will have an impact on inclusion to the PKAS, as described in Table 1

Analysis sets.

#### **5.5** Definition of baseline

Baseline will be defined as the last non-missing data collection point prior to administration of IMP (i.e., linaprazan glurate in Part I) and midazolam (Part II).

## 5.6 Rounding principles

Generally, no rounding of data will be done prior to calculating statistics. However, if reported data contains more than 8 significant digits it will be rounded to 8 significant digits in the database.

In statistical output and descriptive summaries, the following principles will be followed:

- Data will be presented as reported in input data in listings.
- 2 significant digits will be used for percentages (for example relative change from baseline).
- p-values and similar statistical output will be presented using 4 decimal points.
- 3 significant digits will be used for PK parameters and similar when presenting min and max values in tables.
- Descriptive summaries of PK parameters and similar (e.g. mean, SD, median etc.) will be presented with 4 significant digits.
- Descriptive summaries of all other numerical data (e.g. mean, SD, median etc.) will be presented with one extra decimal compared to reported input data.

#### 5.7 Significance level

All statistical hypotheses in this study will be answered using two-sided 90% confidence intervals. This is not a confirmatory study. Hence, point estimates and CIs will be used exploratorily.

## 5.8 Multiple comparisons/multiplicity

No adjustment for multiple comparison/multiplicity will be performed. All significant findings will be reviewed for medical relevance

#### 5.9 Handling of dropouts, missing data and outliers

Outliers will be included in summary tables and listings and will not be handled separately in any analyses. Generally, no imputation of data will be performed. However, when calculating statistics for PK plasma concentrations, concentrations under LLOQ will be replaced with LLOQ/2 if more than 50% of the values for a given time point is above LLOQ. Otherwise, no






statistics will be calculated for that time point. For imputation of PK plasma concentration below LLOQ with the purpose of calculating PK parameters, see Section 9 below.

In case of missing start and stop times of AEs that cannot be investigated further, missing data will be imputed according to a worst-case scenario. This means that start time will be imputed as the closest time point post first intake of IMP and end time as 23:59, resulting in the longest possible treatment emergent duration of the AE.




# 6 CHANGES FROM THE CLINICAL STUDY PROTOCOL

NA




#### 7 CLINICAL DATABASE PROCESSING

#### 7.1 General information

The clinical database is processed and generated according to The Clinical Data Interchange Standards Consortium (CDISC). CDISC is a Standard Developing Organization which develops and publishes standards to normalise the structure of clinical study data and thereby simplify submissions to and reviews by authorities such as the Food and Drug Administration (FDA).

The CDISC standards for clinical studies are the Study Data Tabulation Model (SDTM) and the Analysis Data Model (ADaM). The study data will be structured into a database model reflecting the SDTM and be compliant to SDTM Implementation Guide (SDTM-IG) version 3.2. The data used for statistical analysis will be structured to reflect the Analysis Data Model (ADaM) and be compliant to ADaM Implementation Guide (ADaM-IG) version 1.1.

Data values are collected according to, or mapped into, Controlled Terminology (CT) codelists defined by CDISC, whenever possible. The codelists are updated quarterly at CTC and the latest version available at study start will be used. As per default, CT codelists will be used in all tables, listings, and figures. Custom codelists for test or parameter names will be used if applicable upon Sponsor's request, to align with protocol texts, or to adhere to other standard naming conventions (e.g. PK parameter name "Tmax" will be used instead of the CDISC term "Time of CMAX"). These custom codelists will be mapped in the "Parameter Name" field in the ADaM structure, while the CT will be kept in the SDTM predecessor fields to provide traceability back to CDISC codelists.

### 7.1.1 CDISC Compliance

The study database will be CDISC compliant which means that the clinical database will be processed and generated according to CDISC standard. The database will be validated against SDTM and ADaM Validation rules using Pinnacle 21.

The following CDISC documentation will be generated:

- SDTM Data Definition Specification (also referred to as a Define -XML)
  - Define-XML transmits metadata that describes any tabular dataset structure and supports the interchange of dataset metadata for clinical research applications in a machine-readable format.
- ADaM Data Definition Specification (also referred to as a Define -XML)
  - Define-XML transmits metadata that describes any tabular dataset structure and supports the interchange of dataset metadata for clinical research applications in a machine-readable format.
- Annotated eCRF
  - Links the data collection fields used to capture study data to the corresponding variables in the study database. It enables the user to understand how the study data were collected and to trace back from study analysis results to the origin where it was collected.
- SDTM Reviewers' Guide
  - Intended to provide additional context and act as a single point of orientation for the SDTM datasets.
- ADaM Reviewers' Guide
  - Provides regulatory agency reviewers an orientation to the submitted analysis data in a consistent way and usable format.




### 7.2 Database modeling of study design

The study design is mapped to a SDTM study design model containing the following structural components:

**EPOCH**: An interval of time in the planned conduct of a study. An epoch is associated with a purpose (e.g., screening, randomization, treatment, follow-up), and applies across all arms of the study. Study epochs follow a controlled terminology to represent the different study parts (e.g. SCREENING, TREATMENT [X], FOLLOW-UP)

**ELEMENT**: Building blocks used to build up the entire study length for all subjects. Information on ELEMENTs is extracted from the study design and schedule of events in the protocol. ELEMENTs are defined to span the entire study without gaps. One EPOCH may contain one or several ELEMENTs. All ELEMENTs must have transition rules in accordance with the protocol to determine start and end.

**ARM**: Subjects are allocated to study arms depending on the study design, either by randomization or other allocation processes defined in the study protocol. ARMs are defined as the total number of planned ways a subject can go through the study (unique combination of study ELEMENTs). All ARMs must contain a unique sequence of ELEMENTs.

**VISIT**: Study visits are defined as planned timepoints during the study where study data is collected. A visit can be performed in clinic, by off-site contact with study personnel (phone call, video conference or similar), or by subject initiated recordings of data. The visit schedule is extracted from protocol and eCRF design.

A schematic representation of the SDTM study design is presented in Figure 1.

Figure 1 Schematic representation of the SDTM study design

#### Part I:



<sup>\*</sup>End of study is modeled as a unique visit, but it is performed together with the last participation in the study.

#### Part II:



<sup>\*</sup>End of study is modeled as a unique visit, but it is performed together with the last participation in the study.




## 8 STATISTICAL DELIVERABLES

The following items will be delivered:

- Statistical analyses, summary tables, listings and figures as described under Section 10.
- Clinical study database delivered as a SAS-export file.
- Define -XML for SDTM
- Define -XML for ADaM
- Annotated eCRF
- SDTM Reviewer's Guide
- ADaM Reviewer's Guide




#### 9 STATISTICAL METHODOLOGY

There will be two clean files (CF) in this study, corresponding to the two study parts. Therefore, output in this study (tables, figures and listings) will be done in two different sets, one per study part. However, there will only be one CSR including both study parts.

All collected data will be listed by treatment and subject.

Details on statistical analyses and descriptive summaries are specified below.

All statistical analysis and descriptive summaries will be performed using SAS version 9.4 (SAS institute, Cary, NC).

#### 9.1 Pharmacokinetic calculations

PK parameters will be calculated by Non-Compartmental Analysis (NCA) using the software Phoenix WinNonlin<sup>®</sup> version 8.3 (Certara, U.S.A).

The following NCA PK parameters will be calculated for linaprazan glurate and linaprazan, for secondary endpoints the parameters will only be calculated when feasible:

- C<sub>max</sub> The maximum observed plasma concentration
- AUC<sub>0-t</sub> The area under the plasma concentration versus time curve (AUC) from timepoint 0 to t, where t represents the timepoint of the last detectable plasma concentration per dosing occasion.
- Partial AUCs- AUC from time t<sub>1</sub> to time t<sub>2</sub>. Partial AUCs will be calculated between 0-24 h, 24-48 h Day 2 and 0-24 h Day 14 (only in Part II)
- AUC<sub>0-inf</sub> AUC from timepoint 0 extrapolated to infinity (not calculated for steady state/repeated dose data)
- AUC<sub>tau</sub> AUC per dosing interval (calculated at steady state and for the first dose)
- T<sub>max</sub> Time to reach C<sub>max</sub>
- CL/F Total body clearance for extravascular administration (only for linaprazan glurate as there is no dose data for linaprazan)
- $V_z/F$  Apparent volume of distribution associated with terminal slope (only for linaprazan glurate as there is no dose data for linaprazan)
- $T_{1/2}$  The terminal plasma elimination half-life
- AUC<sub>extr%</sub> Percentage of AUC<sub>0-inf</sub> due to extrapolation from T<sub>last</sub> to infinity
- $R_{acc} C_{max}$  Accumulation ratio for  $C_{max}$  (only in Part II)
- R<sub>acc</sub> AUC Accumulation ratio for AUC (only in Part II)

The following NCA PK parameters will be calculated for clarithromycin:

- AUC<sub>tau</sub> The AUC during dosing interval at steady state
- C<sub>max</sub>
- T<sub>max</sub>
- T<sub>1/2</sub>

The following NCA PK parameters will be calculated for midazolam:

- AUC<sub>0-t</sub>
- AUC<sub>0-inf</sub>
- AUC<sub>extr</sub>%




- C<sub>max</sub>
- T<sub>max</sub>
- $T_{1/2}$
- CL/F
- V<sub>z</sub>/F

Additional PK parameters that will be calculated (and only presented in listing if not specified above) for linaprazan glurate, linaprazan, clarithromycin and midazolam:

- Lambda<sub>z</sub> The eliminate rate constant associated with the terminal phase of the curve
- Rsq adj Coefficient of determination adjusted for the independent variable time
- No points lambda<sub>z</sub> Number of points used in computing lambda<sub>z</sub>
- Lambda<sub>z</sub> lower Lower limit on time included in the calculation of lambda<sub>z</sub>
- Lambda<sub>z</sub> upper Upper limit on time included in the calculation of lambda<sub>z</sub>
- Span The ratio between the interval used for determination of lambda<sub>z</sub> and the terminal  $T_{1/2}$
- AUC<sub>extr</sub>%

Non-compartmental analysis will be based on the actual sampling times recorded during the study. For the purpose of calculating PK parameters, concentrations below lower limit of quantification (LLOQ) occurring before  $C_{max}$  will be treated as zero. Concentrations below LLOQ occurring after  $C_{max}$  will be omitted from the analysis.

 $T_{max}$  and  $C_{max}$  will be based on the observed plasma concentration data.

All AUCs will be assessed by integration of the plasma concentration vs time curve using linear interpolation for increasing plasma levels and logarithmic interpolation for decreasing plasma levels (Linear Up-Log Down method using uniform weighting).

 $AUC_{0-t}$  will be calculated from time 0 to the time t of the last detectable plasma concentration. For  $AUC_{0-inf}$  the area will be calculated to the last timepoint showing a measurable plasma concentration and then extrapolated to infinity using the concentration in the last quantifiable sample and lambda<sub>z</sub>.

$$AUC_{0-inf} = AUC_{0-t} + \frac{C_{last}}{lambda_z}$$

Partial AUC (possible relevant for AUC<sub>tau</sub> calculations) will be derived according to specified time windows, if the end time of the interval does not occur at an actual timepoint either linear interpolation or extrapolation will be used for derivation of the partial AUC. Extrapolation, using lambda<sub>z</sub>, will only be used if the end time of specified interval occur after last detectable plasma concentration.

Formulas for calculation of AUC

• Linear trapezoidal rule:

$$AUC|_{t1}^{t2} = \delta t \times \frac{C_1 + C_2}{2}$$

• Logarithmic trapezoidal rule:




Statistical Analysis Plan for Part I and Part II CX842A2105 FINAL v1.0

astical Analysis Plan for Part I and 
$$AUC|_{t1}^{t2} = \delta t \times \frac{C_2 - C_1}{\ln{\frac{C_2}{C_1}}}$$

where t = time, c = concentration,  $\delta t = t_2 - t_1$ .

Formulas for interpolation (to find C\* at time t\* for  $t1 < t^* < t2$ )

• Linear interpolation rule:

$$C^* = C_1 + \left| \frac{t^* - t_1}{t_2 - t_1} \right| (C_2 - C_1)$$

• Logarithmic interpolation rule:

$$C^* = exp(ln(C_1) + |\frac{t^* - t_1}{t_2 - t_1}| * (ln(C_2) - ln(C_1)))$$

where t = time, c = concentration

Lambda<sub>z</sub>, the first order rate constant associated with the terminal portion of the curve, will be determined by lin-logarithmic regression of the terminal elimination phase of individual plasma concentration vs time curves. Determination of lambda<sub>z</sub> requires identification of a sufficiently linear terminal phase (as determined by visual inspection of the lin-log plasma concentration vs time plot with the regression line) consisting of at least 3 terminal concentration values (not including  $C_{max}$ ). If this is not achieved, lambda<sub>z</sub> and its dependent PK parameters will not be reported for that profile.

In the following cases, lambda $_z$  dependent PK parameters will be flagged in listings as potentially unreliable:

- Lambda<sub>z</sub> estimation is based on a period of less than 1.5 times the resulting  $T_{\frac{1}{2}}$ .
- The adjusted  $R_2$  value of the regression line is < 0.85.
- The estimated % extrapolated AUC is  $\geq 20\%$  ((AUC<sub>0-inf</sub>-AUC<sub>0-last</sub> / AUC<sub>0-inf</sub>)\*100).
  - o In case the extrapolated AUC is > 30% lambda<sub>z</sub> dependent parameter will excluded from analysis and descriptive statistics.

 $T_{1/2}$  will be calculated by ln2 /  $lambda_z$ , and Span will be calculated by  $(lambda_z\_upper - lambda_z\_lower)$  /  $T_{1/2}$ .

CL/F for single doses will be calculated by Dose /  $AUC_{0-inf}$  and CL/F at steady state will be calculated by Dose /  $AUC_{tau}$ .

 $V_z/F$  for single doses will be calculated by Dose / (lambda<sub>z</sub> x AUC<sub>0-inf</sub>), and  $V_z/F$  at steady state will be calculated by Dose / (lambda<sub>z</sub> x AUC<sub>tau</sub>).

The accumulation ratio for  $C_{max}$  will be calculated by  $C_{max}$  at steady state /  $C_{max}$  first dose, and the accumulation ratio for AUC will be calculated by AUC<sub>tau</sub> at steady state / AUC<sub>tau</sub> first dose.




If there is a confirmed dosing error during the study, the pharmacokinetic data for that period will only be included in the listings but excluded from descriptive and statistical analyses. In case of missed blood samples, potential impact on PK parameters will be assessed for each individual case. PK parameters with a high degree of uncertainty due to missing samples (e.g. multiple samples missing around  $C_{max}$ ) will be flagged as unreliable in the report and may in rare cases be excluded from summary tables, descriptive statistics, and statistical analysis.

Relevant PK data will be presented by using summary statistics with number of measurements, arithmetic mean, SD, as well as median, minimum and maximum values. In addition, for the parameters AUC and  $C_{max}$  the geometric mean and coefficient of variation (CV%) will be presented.

## 9.2 Analysis of the primary endpoint

## 9.2.1 Analysis of PK parameters

#### Part I:

The following PK parameters will be assessed for linaprazan glurate and linaprazan, in the presence (Day 10) and absence (Day 1) of clarithromycin administration:

- AUC<sub>0-inf</sub>
- AUC<sub>0-t</sub>
- C<sub>max</sub>

#### Part II:

The following PK parameters will be assessed for midazolam, in the presence (Day2 and 14 respectively) and absence (Day 1) of linaprazan glurate administration:

- AUC<sub>0-inf</sub>
- AUC<sub>0-t</sub>
- C<sub>max</sub>

## 9.2.2 Mixed model for PK parameters Part I

The PK parameters  $AUC_{inf}$ ,  $AUC_{0-t}$  and  $C_{max}$  will be analyzed using a mixed model following a natural logarithmic transformation, with fixed effect for treatment and random effect for subject. Kenward-Rogers approximation for degrees of freedom will be used. Model results will be back-transformed to the original scale to present, ratios of geometric means together with 2-sided 90% CI of test treatment (linaprazan glurate + clarithromycin) and reference treatment (linaprazan glurate alone) will be estimated and presented. The same analysis will also be done for linaprazan + clarithromycin vs. linaprazan alone. The SAS proc mixed code to be used will be:




## 9.2.3 Mixed model for PK parameters Part II

Midazolam PK parameters  $AUC_{inf}$ ,  $AUC_{0-t}$  and  $C_{max}$  for the comparisons midazolam + linaprazan glurate Day 14 / midazolam Day 1, midazolam + linaprazan glurate Day 14 / midazolam + linaprazan glurate Day 2 and midazolam + linaprazan glurate Day 2 / midazolam Day 1 will be estimated using the same model as described under section 9.2.2 above.

## 9.3 Analysis of secondary endpoints

#### 9.3.1 Adverse events

An overview of all AEs, including SAEs, intensity, relationship to IMP, and deaths will be presented. The incidence of AEs and SAEs will be summarized by SOC and PT by treatment and overall. An overview of any treatment-related AEs will be summarized by SOC and PT if considered appropriate.

### 9.3.2 Physical examinations

Clinically significant and non-clinically significant abnormal findings will be specified and presented by subject and summarized by treatment.

#### 9.3.3 Vital signs

Vital signs (systolic/diastolic BP, pulse rate, and body temperature) will be summarized by treatment and overall. Data will be presented with absolute and percent change from baseline.

### 9.3.4 12-lead safety ECG

All ECGs will be categorized as "normal", "abnormal, not clinically significant", or "abnormal, clinically significant" (as judged by the Investigator) and summarized by treatment using frequency tables.

#### 9.3.5 Safety laboratory analyses

Safety laboratory data will be summarized by treatment, with absolute and percent change from baseline at each visit.

Abnormal, clinically significant values will be summarized separately if considered appropriate.

# 9.3.6 Additional PK parameters Part I for linaprazan glurate and linaprazan, not limited to:

The following secondary NCA PK parameters will be assessed for linaprazan glurate and linaprazan, but are not limited to:

- T<sub>max</sub>
- $T_{1/2}$
- CL/F
- V/F
- AUCextr%




# 9.3.7 Clarithromycin PK parameters Part I with and without co-administration of linaprazan glurate:

The following secondary NCA PK parameters will be assessed for clarithromycin with and without co-administration of linaprazan glurate, not limited to:

- AUC to the end of the dosing period (AUC<sub>tau</sub>)
- C<sub>max</sub>
- T<sub>max</sub>
- $T_{1/2}$

# 9.3.8 Additional Midazolam PK parameters Part II in the presence and absence of linaprazan glurate administration (if feasible):

The following secondary NCA PK parameters will be assessed for midazolam, in the presence and absence of linaprazan glurate administration (if feasible):

- T<sub>max</sub>
- T<sub>1/2</sub>
- AUCextr%
- CL/F
- V/F

## 9.3.9 Linaprazan glurate and linaprazan PK parameters Part II (if feasible):

The following secondary NCA PK parameters will be assessed for linaprazan glurate and linaprazan (if feasible):

- AUC<sub>tau</sub>
- AUC<sub>0-t</sub>
- C<sub>max</sub>
- AUC<sub>extr</sub>%
- CL/F (only for linaprazan glurate)
- V/F (only for linaprazan glurate)
- Racc
- T<sub>max</sub>
- T<sub>1/2</sub>

Additional PK parameters may be determined if deemed appropriate.

## 9.4 Description of study population

Other study population/demographics data will be presented in listings and summarized descriptively as described in section 10 below.




## 10 DATA DISPLAY PLAN

| 10.1 | Tal | ble of contents DDP | |
|---|---|---|---|
| 10.2 | Stu | udy tables | . 27 |
| 10.2 | 2.1 | Demographic data | . 27 |
| 10.2 | 2.2 | Primary endpoints | . 32 |
| 1 | 0.2. | 2.1 Analysis of pharmacokinetics | . 32 |
| 10.2 | 2.3 | Secondary endpoints | . 36 |
| 1 | 0.2. | 3.1 Additional PK parameters Part I | . 36 |
| 1 | 0.2. | 3.2 Additional PK parameters Part II | . 38 |
| 1 | 0.2. | 3.3 Adverse events | . 41 |
| 1 | 0.2. | 3.4 Physical examinations | . 43 |
| 1 | 0.2. | 3.5 Vital signs | . 44 |
| 1 | 0.2. | 3.6 12-lead safety ECG | . 45 |
| 1 | 0.2. | 3.7 Safety laboratory analyses | . 45 |
| 10.3 | Stu | ıdy figures | . 46 |
| 10 | <i>3.1</i> | Primary endpoint(s) | . 46 |
| 10.4 | Stu | ıdy listings | . 48 |
| List of t | able | s | |
| Table Di | M 1 | Baseline characteristics and demographics for Part I (Full analysis set) | 27 |
| Table Di | M 2 | Baseline characteristics and demographics for Part II (Full analysis set) | 28 |
| Table DS | S 1 | Subject disposition for Part I (All subjects) | 29 |
| Table DS | S 2 | Subject disposition for Part II (All subjects) | 30 |
| Table M analysis | | Medical history events by system organ class and preferred term part I (Fu 30 | ıll |
| Table M analysis | | Medical history events by system organ class and preferred term part II (F 30 | ull |
| Table Cl | M 1 | Prior medications by ATC levels 4 and 5 for Part I (Full analysis set) | 31 |
| Table Cl | M 2 | Prior medications by ATC levels 4 and 5 for Part II (Full analysis set) | 31 |
| Table CN set) | М 3 | Concomitant medications by ATC levels 4 and 5 for Part I (Full analysis 31 | |
| Table CN set) | M 4 | Concomitant medications by ATC levels 4 and 5 for Part II (Full analysis 31 | |




| Table PP 1 (Pharmacokinet | PK parameters for linaprazan glurate and linaprazan for Part I tic analysis set) | 32 |
|---|---|---|
| Table PP 2 | PK parameters for midazolam for Part II (Pharmacokinetic analysis set) | 33 |
| Table PP 3 set) | Mixed model results for PK parameters for Part I (Pharmacokinetic analy 34 | 'sis |
| Table PP 4 set) | Mixed model results for PK parameters for Part II (Pharmacokinetic anal 34 | ysis |
| Table PP 5<br>(Pharmacokinet | Additional PK parameters for linaprazan glurate and linaprazan for Part litic analysis set) | 36 |
| Table PP 6 set) | PK parameters for clarithromycin for Part I (Pharmacokinetic analysis 37 | |
| Table PP 7 analysis set) | Additional PK parameters for midazolam for Part II (Pharmacokinetic 38 | |
| Table PP 8<br>(Pharmacokine | Additional PK parameters for linaprazan glurate and linaprazan for Part I tic analysis set) | II<br>39 |
| Table PC 1 | Plasma concentrations for part I (Pharmacokinetic analysis set) | 35 |
| Table PC 2 | Plasma concentrations for part II (Pharmacokinetic analysis set) | 35 |
| Table AE 1 | Overview of adverse events for Part I (Full analysis set) | 41 |
| Table AE 2 | Overview of adverse events for Part II (Full analysis set) | 41 |
| Table AE 3 analysis set) | Adverse events by system organ class and preferred term for Part I (Full 42 | |
| Table AE 4 analysis set) | Adverse events by system organ class and preferred term for Part II (Full 42 | |
| Table PE 1 | Physical examinations for Part I (Full analysis set) | 43 |
| Table PE 2 | Physical examinations for Part II (Full analysis set) | 43 |
| Table VS 1 | Vital signs measurements for Part I (Full analysis set) | 44 |
| Table VS 2 | Vital signs measurements for Part II (Full analysis set) | 44 |
| Table EG 1 | ECG measurements for Part I (Full analysis set) | 45 |
| Table EG 2 | ECG measurements for Part II (Full analysis set) | 45 |
| Table EG 3 | ECG interpretations for Part I (Full analysis set) | 45 |
| Table EG 4 | ECG interpretations for Part II (Full analysis set) | 45 |




| • | Statistical Alialysis Flatt 1 and Fatt 11 CA642A2103 FINAL VI.0 |
|---|---|
| Table LB 1 set) | Safety laboratory measurements - clinical chemistry for part I (Full analysis 45 |
| Table LB 2 set) | Safety laboratory measurements - clinical chemistry for part II (Full analysis $45$ |
| Table LB 3 set) | Safety laboratory measurements - haematology for part I (Full analysis 45 |
| Table LB 4 set) | Safety laboratory measurements - haematology for part II (Full analysis 45 |
| Table LB 5 | Safety laboratory interpretations – urinalysis for part I (Full analysis set) 45 |
| Table LB 6 | Safety laboratory interpretations – urinalysis for part II (Full analysis set) 45 |
| List of figures | |
| Figure PC 1 (Pharmacokinetic | Geometric mean plasma concentrations over time (lin-log) for Part I analysis set) 46 |
| Figure PC 2 (Pharmacokinetic | Geometric mean plasma concentrations over time (lin-log) for Part II analysis set) 46 |
| Figure PC 3 (Pharmacokinetic | Geometric mean plasma concentrations over time (lin-lin) for Part I analysis set) 46 |
| Figure PC 4 (Pharmacokinetic | Geometric mean plasma concentrations over time (lin-lin) for Part II analysis set) 46 |
| Figure PC 5 set) | Individual plasma concentrations over time (lin-log) for Part I (Full analysis 47 |
| Figure PC 6 set) | Individual plasma concentrations over time (lin-log) for Part II (Full analysis 47 |
| Figure PC 7 set) | Individual plasma concentrations over time (lin-lin) for Part I (Full analysis 47 |
| Figure PC 8 | Individual plasma concentrations over time (lin-lin) for Part II (Full analysis 47 |




## 10.2 Study tables

## 10.2.1 Demographic data

# Table DM 1 Baseline characteristics and demographics for Part I (Full analysis set)

| Assessment (unit) | | Total<br>(N=XX) |
|---|---|---|
| Age (years) | n | x |
| | Mean (SD) | xx.x (xx.x) |
| | Median (Min, Max) | xx.x (xx, xx) |
| Height (cm) | n | x |
| | Mean (SD) | xxx.x (xx.x) |
| | Median (Min, Max) | xxx.x (xxx, xxx) |
| Weight (kg) | n | x |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) |
| Body Mass Index (kg/m2) | n | X |
| | Mean (SD) | xx.xx (xx.xx) |
| | Median (Min, Max) | xx.xx (xx.x, xx.x) |
| Sex | Female | xx (xx%) |
| | Male | xx (xx%) |
| Ethnicity | Hispanic or latino | xx (xx%) |
| | Not hispanic or latino | xx (xx%) |
| | Not reported | xx (xx%) |
| | Unknown | xx (xx%) |
| Race | American Indian or Alaska Native | xx (xx%) |
| | Asian | xx (xx%) |
| | Black or African American | xx (xx%) |
| | Native Hawaiian or Other Pacific Islander | xx (xx%) |




## Statistical Analysis Plan for Part I and Part II CX842A2105 FINAL v1.0

| Assessment (unit) | | Total<br>(N=XX) |
|-------------------|-------|-----------------|
| | White | xx (xx%) |

Data based on [ANALYSIS SET]. N: number of subjects in treatment group. Mean values and percentages are based on n. n: Number of observations. SD: Standard deviation. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

## Table DM 2 Baseline characteristics and demographics for Part II (Full analysis set)

Use the same format as for Table DM 1.




## **Table DS 1** Subject disposition for Part I (All subjects)

| | Total<br>(N=XXX) |
|-----------------------------------------|------------------|
| Screened subjects | xxx |
| Withdrawn prior to dose | xxx |
| Reason for withdrawal prior to dose | |
| Reason 1 | xxx |
| Reason 2 | xxx |
| <del></del> | xxx |
| Subjects included in study | xxx |
| Withdrawn subjects | |
| Reason 1 | xxx |
| Reason 2 | xxx |
| <del></del> | xxx |
| Subjects completing all study visits | xxx |
| ncluded in Full analysis set | xxx |
| ncluded in Pharmacokinetic analysis set | xxx |
| Subjects at each visit | |
| Visit 1 | xxx |
| Visit 2 | xxx |
| Visit 3 | xxx |
| Visit 4 | xxx |
| Visit 5 | xxx |
| Visit 6 | xxx |
| Visit 7 | xxx |
| Visit 8 | xxx |
| Visit 9 | xxx |
| Visit 10 | XXX |

Data based on All subjects. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS




## Table DS 2 Subject disposition for Part II (All subjects)

Use the same format as for Table DS 1

Table MH 1 Medical history events by system organ class and preferred term part I (Full analysis set)

| | Total<br>(N=XX) | |
|-----------------------------------|-----------------|----|
| System organ class Preferred term | n (%) | m |
| Total | xx (xx%) | XX |
| [SOC 1] | xx (xx%) | XX |
| [SOC 1 PT 1] | xx (xx%) | xx |
| [SOC 1 PT 2] | xx (xx%) | XX |
| [SOC 1 PT] | xx (xx%) | XX |
| [SOC 2] | xx (xx%) | XX |
| [SOC 2 PT 1] | xx (xx%) | XX |
| [SOC 2 PT 2] | xx (xx%) | XX |
| [SOC 2 PT] | xx (xx%) | XX |
| [SOC] | xx (xx%) | XX |
| [SOC PT 1] | xx (xx%) | XX |
| [SOC PT 2] | xx (xx%) | XX |
| [SOC PT] | xx (xx%) | XX |

Data based on [ANALYSIS SET]. n, number of subjects. m, number of events. Percentages are based on the number of subjects in the treatment period. The following events are coded with multiple terms and are represented as separate events in tables and listings: '[MH TERM 1], [MH TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

## Table MH 2 Medical history events by system organ class and preferred term part II (Full analysis set)

Use the same format as for Table MH 1.




## Table CM 1 Prior medications by ATC levels 4 and 5 for Part I (Full analysis set)

| | Total<br>(N=XX) | |
|---------------------------------------|-----------------|----|
| ATC classification Active ingredients | n (%) | m |
| Total | xx (xx%) | XX |
| [L4 1] | xx (xx%) | XX |
| [L4 1 L5 1] | xx (xx%) | XX |
| [L4 1 L5 2] | xx (xx%) | XX |
| [L4 1 L5] | xx (xx%) | XX |
| [L4 2] | xx (xx%) | XX |
| [L4 2 L5 1] | xx (xx%) | XX |
| [L4 2 L5 2] | xx (xx%) | XX |
| [L4 2 L5] | xx (xx%) | XX |
| [L4] | xx (xx%) | XX |
| [L4 L5 1] | xx (xx%) | XX |
| [L4 L5 2] | xx (xx%) | XX |
| [L4 L5] | xx (xx%) | XX |

Data based on [ANALYSIS SET]. n, number of subjects. m, number of events. Percentages are based on the number of subjects in the treatment period. The following records are coded with multiple terms and are represented as separate events in tables and listings: '[CM TERM 1], [CM TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

## Table CM 2 Prior medications by ATC levels 4 and 5 for Part II (Full analysis set)

Use the same format as for Table CM 1.

## Table CM 3 Concomitant medications by ATC levels 4 and 5 for Part I (Full analysis set)

Use the same format as for Table CM 1.

## Table CM 4 Concomitant medications by ATC levels 4 and 5 for Part II (Full analysis set)

Use the same format as for Table CM 1.




## 10.2.2 Primary endpoints

## 10.2.2.1 Analysis of pharmacokinetics

Table PP 1 PK parameters for linaprazan glurate and linaprazan for Part I (Pharmacokinetic analysis set)

| Assessment (unit) | | Linaprazan glurate<br>alone<br>(N=XX) | Linaprazan glurate co-<br>administred with<br>clarithromycin<br>(N=XX) | Linaprazan alone<br>(N=XX) | Linaprazan co-<br>administred with<br>clarithromycin<br>(N=XX) |
|---|---|---|---|---|---|
| AUC <sub>inf</sub> (unit) | n | xx | xx | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| AUC <sub>0-t</sub> (unit) | n | xx | xx | xx | xx |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| C <sub>max</sub> (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |

Data based on [population]. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS




## Table PP 2 PK parameters for midazolam for Part II (Pharmacokinetic analysis set)

| Assessment (unit) | | Midazolam alone,<br>Day 1<br>(N=XX) | Midazolam co-<br>administred with<br>linaprazan glurate, Day 2<br>(N=XX) | Midazolam co-<br>administred with<br>2 linaprazan glurate, Day 14<br>(N=XX) |
|---|---|---|---|---|
| AUC <sub>inf</sub> (unit) | n | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| AUC <sub>0-t</sub> (unit) | n | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| C <sub>max</sub> (unit) | n | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |

Data based on [population]. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS


#### Statistical Analysis Plan for Part I and Part II CX842A2105 FINAL v1.0

Table PP 3 Mixed model results for PK parameters for Part I (Pharmacokinetic analysis set)

| Parameter | Test treatment | Reference treatment | 90% CI<br>lower bound | Ratio of geometric least square means | 90% CI<br>upper bound |
|---|---|---|---|---|---|
| AUC <sub>inf</sub> (unit) | Linaprazan glurate co-administred with clarithromycin | Linaprazan glurate alone | X.XXX | x.xxxx | X.XXX |
| | Linaprazan co-administred with clarithromycin | Linaprazan glurate alone | X.XXX | X.XXXX | X.XXX |
| $AUC_{0-t}$ (unit) | Linaprazan glurate co-administred with clarithromycin | Linaprazan glurate alone | x.xxx | X.XXXX | X.XXX |
| | Linaprazan co-administred with clarithromycin | Linaprazan glurate alone | x.xxx | X.XXXX | X.XXX |
| C <sub>max</sub> (unit) | Linaprazan glurate co-administred with clarithromycin | Linaprazan glurate alone | X.XXX | x.xxxx | X.XXX |
| | Linaprazan co-administred with clarithromycin | Linaprazan glurate alone | x.xxx | X.XXXX | x.xxx |

Pairwise treatment comparisons are based on a mixed effects model with treatment as a fixed effect and subject as a random effect. Kenward-Rogers approximation for degrees of freedom has been used.

Data based on PK analysis set.

[STUDYID], SAS program: [PROGRAM NAME]. Run by: [USERNAME], [USER EMAIL] [TIMESTAMP]. Data extracted at: [TIMESTAMP]

Table PP 4 Mixed model results for PK parameters for Part II (Pharmacokinetic analysis set)

| Parameter | Test treatment | Reference treatment | 90% CI<br>lower bound | Ratio of geometric least square means | 90% CI<br>upper bound |
|---|---|---|---|---|---|
| AUC <sub>inf</sub> (unit) | Midazolam co-administred with linaprazan glurate, Day 14 | Midazolam alone, Day 1 | X.XXX | x.xxxx | X.XXX |
| | Midazolam co-administred with linaprazan glurate, Day 2 | Midazolam alone, Day 1 | X.XXX | x.xxxx | X.XXX |
| | Midazolam co-administred with linaprazan glurate, Day 14 | Midazolam co-administred with linaprazan glurate, Day 2 | X.XXX | x.xxxx | X.XXX |
| AUC <sub>0-t</sub> (unit) | Midazolam co-administred with linaprazan glurate, Day 14 | Midazolam alone, Day 1 | X.XXX | x.xxxx | X.XXX |
| | Midazolam co-administred with linaprazan glurate, Day 2 | Midazolam alone, Day 1 | X.XXX | x.xxxx | X.XXX |
| | Midazolam co-administred with linaprazan glurate, Day 14 | Midazolam co-administred with linaprazan glurate, Day 2 | X.XXX | x.xxxx | X.XXX |
| C <sub>max</sub> (unit) | Midazolam co-administred with linaprazan glurate, Day 14 | Midazolam alone, Day 1 | X.XXX | x.xxxx | X.XXX |
| | Midazolam co-administred with linaprazan glurate, Day 2 | Midazolam alone, Day 1 | X.XXX | x.xxxx | X.XXX |
| | Midazolam co-administred with linaprazan glurate, Day 14 | Midazolam co-administred with linaprazan glurate, Day 2 | X.XXX | x.xxxx | x.xxx |

Pairwise treatment comparisons are based on a mixed effects model with treatment as a fixed effect and subject as a random effect. Kenward-Rogers approximation for degrees of freedom has been used.

Data based on PK analysis set.

[STUDYID], SAS program: [PROGRAM NAME]. Run by: [USERNAME], [USER EMAIL] [TIMESTAMP]. Data extracted at: [TIMESTAMP]


## Statistical Analysis Plan for Part I and Part II CX842A2105 FINAL v1.0

## Table PC 1 Plasma concentrations for part I (Pharmacokinetic analysis set)

| Assessment (unit) | Assessment timepoint | | Total<br>(N=XX) |
|---|---|---|---|
| [PARAMETER 1] (unit) | [Assessment timepoint 1] | n | xx |
| | | Mean (SD) | x.xx (x.xx) |
| | | Median (Min, Max) | x.xx(x.x, x.x) |
| | [Assessment timepoint 2] | n | xx |
| | | Mean (SD) | x.xx (x.xx) |
| | | Median (Min, Max) | x.xx (x.x, x.x) |

Data based on [population]. Dynamic footnote based on table content: n: Number of observations. SD: Standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

## Table PC 2 Plasma concentrations for part II (Pharmacokinetic analysis set)

Use the same format as for

Table PC 1.



### 10.2.3 Secondary endpoints

## 10.2.3.1 Additional PK parameters Part I

Table PP 5 Additional PK parameters for linaprazan glurate and linaprazan for Part I (Pharmacokinetic analysis set)

| Assessment (unit) | | Linaprazan glurate<br>alone<br>(N=XX) | Linaprazan glurate co-<br>administred with<br>clarithromycin<br>(N=XX) | Linaprazan alone<br>(N=XX) | Linaprazan co-<br>administred with<br>clarithromycin<br>(N=XX) |
|---|---|---|---|---|---|
| [T <sub>max</sub> ] (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| $[T_{1/2}]$ (unit) | n | xx | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| [CL/F] (unit) | n | xx | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| [V/F] (unit) | n | xx | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| $[AUC_{extr\%}](unit)$ | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |

Data based on [population]. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS




## Table PP 6 PK parameters for clarithromycin for Part I (Pharmacokinetic analysis set)

| Assessment (unit) | | Clarithromycin alone (N=XX) | clarithromycin co-administred<br>with linaprazan glurate<br>(N=XX) |
|---|---|---|---|
| [AUC <sub>tau</sub> ] (unit) | n | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) |
| [C <sub>max</sub> ] (unit) | n | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) |
| $\left[T_{max}\right](unit)$ | n | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| $[T_{1/2}]$ (unit) | n | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx (x.x, x.x) |

Data based on [population]. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS




## 10.2.3.2 Additional PK parameters Part II

Table PP 7 Additional PK parameters for midazolam for Part II (Pharmacokinetic analysis set)

| Assessment (unit) | | Midazolam alone,<br>Day 1<br>(N=XX) | Midazolam co-<br>administred with<br>linaprazan glurate, Day 2<br>(N=XX) | Midazolam co-<br>administred with<br>linaprazan glurate, Day 14<br>(N=XX) |
|---|---|---|---|---|
| [T <sub>max</sub> ] (unit) | n | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| $[T_{1/2}]$ (unit) | n | xx | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| [CL/F] (unit) | n | xx | xx | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| [V/F] (unit) | n | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| [AUC <sub>extr%</sub> ] (unit) | n | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |

Data based on [population]. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS




Table PP 8 Additional PK parameters for linaprazan glurate and linaprazan for Part II (Pharmacokinetic analysis set)

| Assessment (unit) | | Linaprazan glurate,<br>Day 2<br>(N=XX) | linaprazan glurate,<br>Day 14<br>(N=XX) | Linaprazan,<br>Day 2<br>(N=XX) | linaprazan,<br>Day 14<br>(N=XX) |
|---|---|---|---|---|---|
| [AUC <sub>inf</sub> ] (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| [AUC <sub>0-t</sub> ] (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| [C <sub>max</sub> ] (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| [AUC <sub>extr%</sub> ] (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| | Geometric Mean (geo CV%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) | x.xxx (x.x%) |
| CL/F] (unit) | n | xx | XX | NC | NC |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | NC | NC |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | NC | NC |
| V/F] (unit) | n | xx | XX | NC | NC |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | NC | NC |
| | Median (Min, Max) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | NC | NC |
| [R <sub>acc</sub> ] (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx (x.x, x.x) | x.xx (x.x, x.x) |




### Statistical Analysis Plan for Part I and Part II CX842A2105 FINAL v1.0

| Assessment (unit) | | Linaprazan glurate,<br>Day 2<br>(N=XX) | linaprazan glurate,<br>Day 14<br>(N=XX) | Linaprazan,<br>Day 2<br>(N=XX) | linaprazan,<br>Day 14<br>(N=XX) |
|---|---|---|---|---|---|
| [T <sub>max</sub> ] (unit) | n | xx | XX | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx(x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |
| $[T_{1/2}]$ (unit) | n | xx | xx | XX | XX |
| | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) | x.xx(x.x, x.x) |

Data based on [population]. n: Number of observations. SD: Standard deviation. CV%: Coefficient of variation described as percentage. Geo CV%: Geometric coefficient of variation described as percentage calculated using log-transformed standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS




### 10.2.3.3 Adverse events

Table AE 1 Overview of adverse events for Part I (Full analysis set)

| | Total<br>(N=XX) | | linaprazan glurate<br>4)<br>(N=XX) | e (Visit 2 to | clarithromycin (V<br>(N=XX) | Visit 5) | linaprazan glurat<br>clarithromycin (V<br>(N=XX) | | Follow-up<br>(N=XX) | |
|---|---|---|---|---|---|---|---|---|---|---|
| | n (%) | m | n (%) | m | n (%) | m | n (%) | m | n (%) | m |
| Any AE | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Any SAE | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Any AE leading to withdrawal from study | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| Any AE leading to death | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Causality | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [Unlikely related] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [Possibly related] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [Probably related] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Severity | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Grade 1 - Mild | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Grade 2 - Moderate | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx |
| Grade 3 - Severe | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Grade 4 - Life-Threatening | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| Grade 5 - Death | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |

AEs are allocated to respective columns, if the AE starts during the time window indicated by the column headings. Data based on [ANALYSIS SET]. N: number of subjects in treatment group. Percentages are based on N. n, number of subjects. m, number of events. The following AEs are coded with multiple MedDRA terms and are represented as separate AEs in tables and listings: '[AE TERM 1]', '[AE TERM 2]', '[AE TERM 3]. See listings for detailed information. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

### Table AE 2 Overview of adverse events for Part II (Full analysis set)

Use the same format as for Table AE 1. Change the column headings to the relevant victim and perpetrator drugs.




Table AE 3 Adverse events by system organ class and preferred term for Part I (Full analysis set)

| Total<br>(N=XX) | | | linaprazan glurate (Visit 2 clarithromycin (Visit 5) to 4) (N=XX) | | | linaprazan glurate and Follow-up clarithromycin (Visit 6 to 9) (N=XX) (N=XX) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| System organ class<br>Preferred term | n (%) | m | n (%) | m | n (%) | m | n (%) | m | n (%) | m |
| Total | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC 1 PT 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT 2] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 1 PT] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx |
| [SOC 2 PT 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX |
| [SOC 2 PT 2] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx |
| [SOC 2 PT] | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | xx |
| [SOC] | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC PT 1] | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC PT 2] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | XX | xx (xx%) | xx |
| [SOC PT] | xx (xx%) | xx | xx (xx%) | xx | xx (xx%) | XX | xx (xx%) | xx | xx (xx%) | XX |

AEs are allocated to respective columns, if the AE starts during the time window indicated by the column headings. Data based on [ANALYSIS SET]. N, number of subjects. M, number of events. Percentages are based on the number of subjects in the treatment period. The following events are coded with multiple terms and are represented as separate events in tables and listings: '[AE TERM 1], [AE TERM 2]'. See listings for detailed information. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

## Table AE 4 Adverse events by system organ class and preferred term for Part II (Full analysis set)

Use the same format as for Table AE 3. Change the column headings to the relevant victim and perpetrator drugs.




## 10.2.3.4 Physical examinations

Table PE 1 Physical examinations for Part I (Full analysis set)

| Assessment | Assessment timepoint | | Total<br>(N=XX) |
|--------------|----------------------|--------------|-----------------|
| PARAMETER 1] | Screening | Normal | x (xx%) |
| | | Abnormal NCS | x (xx%) |
| | | Abnormal CS | x (xx%) |
| | | Not assessed | x (xx%) |
| | Visit 2 | Normal | x (xx%) |
| | | Abnormal NCS | x (xx%) |
| | | Abnormal CS | x (xx%) |
| | | Not assessed | x (xx%) |
| | End of study | Normal | x (xx%) |
| | | Abnormal NCS | x (xx%) |
| | | Abnormal CS | x (xx%) |
| | | Not assessed | x (xx%) |

Data based on [population]. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

## Table PE 2 Physical examinations for Part II (Full analysis set)

Use the same format as for Table PE 1.




### 10.2.3.5 Vital signs

Table VS 1 Vital signs measurements for Part I (Full analysis set)

| Assessment (unit) | Result category | Assessment timepoint | | Total<br>(N=XX) |
|---|---|---|---|---|
| [PARAMETER 1] (unit) | it) Measured value [Assessment timepoint 1] | | n | XX |
| | | | Mean (SD) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) |
| | | [Assessment timepoint 2] | n | XX |
| | | | Mean (SD) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) |
| | Absolute change from baseline | [Assessment timepoint 2] | n | xx |
| | | | Mean (SD) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx(x.x, x.x) |
| | Relative change from baseline (%) | [Assessment timepoint 2] | n | XX |
| | | | Mean (SD) | x.xx (x.xx) |
| | | | Median (Min, Max) | x.xx (x.x, x.x) |

Data based on [population]. Dynamic footnote based on table content: n: Number of observations. SD: Standard deviation. NC: Not calculated - number of evaluable observations less than 3. NA: Not available - no evaluable observations. SAS program: [PROGRAM NAME].sas. Run by: [USERNAME] YYYY-MM-DDTHH:MM:SS. Data extracted at: YYYY-MM-DDTHH:MM:SS

### Table VS 2 Vital signs measurements for Part II (Full analysis set)

Use the same format as for Table VS 1.




### 10.2.3.6 12-lead safety ECG

### Table EG 1 ECG measurements for Part I (Full analysis set)

Use the same format as for Table VS 1.

### Table EG 2 ECG measurements for Part II (Full analysis set)

Use the same format as for Table VS 1.

### Table EG 3 ECG interpretations for Part I (Full analysis set)

Use the same format as for Table PE 1.

### Table EG 4 ECG interpretations for Part II (Full analysis set)

Use the same format as for Table PE 1.

### 10.2.3.7 Safety laboratory analyses

## Table LB 1 Safety laboratory measurements - clinical chemistry for part I (Full analysis set)

Use the same format as for Table VS 1.

## Table LB 2 Safety laboratory measurements - clinical chemistry for part II (Full analysis set)

Use the same format as for Table VS 1.

## Table LB 3 Safety laboratory measurements - haematology for part I (Full analysis set)

Use the same format as for Table VS 1.

## Table LB 4 Safety laboratory measurements - haematology for part II (Full analysis set)

Use the same format as for Table VS 1.

# Table LB 5 Safety laboratory interpretations – urinalysis for part I (Full analysis set) Use the same format as for Table VS 1.

# Table LB 6 Safety laboratory interpretations – urinalysis for part II (Full analysis set) Use the same format as for Table VS 1.




### 10.3 Study figures

### 10.3.1 Primary endpoint(s)

Figure PC 1 Geometric mean plasma concentrations over time (lin-log) for Part I (Pharmacokinetic analysis set)



Data based on [ANALYSIS SET].
[STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: [PROGRAM NAME]. Run by: [USERNAME],
[TIMESTAMP]

Plot all PK profiles in the same graph – Victim drug, perpetrator drug and victim drug + perpetrator drug -> 3 series in the same graph, with a legend outlining which data series corresponds to what (combination of) drugs.

## Figure PC 2 Geometric mean plasma concentrations over time (lin-log) for Part II (Pharmacokinetic analysis set)

Use the same format as for Figure PC 1.

# Figure PC 3 Geometric mean plasma concentrations over time (lin-lin) for Part I (Pharmacokinetic analysis set)

Use the same format as for Figure PC 1, but plot on linear Y-axis scale.

# Figure PC 4 Geometric mean plasma concentrations over time (lin-lin) for Part II (Pharmacokinetic analysis set)

Use the same format as for Figure PC 1, but plot on linear Y-axis scale.




Figure PC 5 Individual plasma concentrations over time (lin-log) for Part I (Full analysis set)



Data based on [ANALYSIS SET].

[STUDYID] [DOMAIN]: [PARAMETER CATEGORY], SAS program: [PROGRAM NAME]. Run by: [USERNAME], [TIMESTAMP]

Plot all PK profiles in the same graph – Victim drug, perpetrator drug and victim drug + perpetrator drug -> 3 series in the same graph, with a legend outlining which data series corresponds to what (combination of) drugs.

# Figure PC 6 Individual plasma concentrations over time (lin-log) for Part II (Full analysis set)

Use the same format as for Figure PC 5.

# Figure PC 7 Individual plasma concentrations over time (lin-lin) for Part I (Full analysis set)

Use the same format as for Figure PC 5, but plot on linear Y-axis scale.

# Figure PC 8 Individual plasma concentrations over time (lin-lin) for Part II (Full analysis set)

Use the same format as for Figure PC 5, but plot on linear Y-axis scale.




### 10.4 Study listings

Produce separate listings for Part I and Part II respectively. Update listings titles to reflect which Part is intended.

### 16.2.1 Discontinued subjects

- Listing 16.2.1-1 Discontinued subjects (All subjects)
- Listing 16.2.1- 2 Non-eligible subjects (All subjects)
- Listing 16.2.1-3 Disposition (All subjects)
- Listing 16.2.1-4 Subject visits (All subjects)
- Listing 16.2.1-5 Subject elements (All subjects)

#### 16.2.2 Protocol deviations

- Listing 16.2.2-1 Protocol deviations (All subjects)
- 16.2.3 Subjects excluded from the efficacy analysis
- Listing 16.2.3-1 Subjects excluded from Full analysis set (All subjects)
- Listing 16.2.3- 2 Subjects excluded from Pharmacokinetic analysis set (All subjects)
- Listing 16.2.3- 3 Population definitions (All subjects)

### 16.2.4 Demographic data

- Listing 16.2.4-1 Demography (Full analysis set)
- Listing 16.2.4- 2 Medical History (Full analysis set)
- Listing 16.2.4-3 Prior and concomitant medications (Full analysis set)

### 16.2.5 Compliance and/or Drug Concentration Data

- Listing 16.2.5-1 Plasma concentration data (Full analysis set)
- Listing 16.2.5-2 Pharmacokinetic parameters (Full analysis set)
- Listing 16.2.5-3 Treatment compliance (Full analysis set)




### 16.2.6 Individual Efficacy Response Data

• Listing 16.2.6-1 IMP administration (Full analysis set)

### 16.2.7 Adverse event listings (each subject)

- Listing 16.2.7-1 Adverse events (Full analysis set)
- Listing 16.2.7-2 Serious adverse events (Full analysis set)

### 16.2.8 Listings of individual laboratory measurements by subject

• Listing 16.2.8-1 Safety laboratory measurements (Full analysis set)

Abnormal values and assessment of clinical significance must be included.

• Listing 16.2.8-2 Other laboratory measurements (Full analysis set)
Urine drug screen, alcohol test, pregnancy test

### 16.2.9 Listings of vital signs, ECG, physical examination data by subject

- Listing 16.2.9-1 Vital signs (Full analysis set)
- Listing 16.2.9-2 ECG (Full analysis set)
- Listing 16.2.9-3 Physical examinations (Full analysis set)
